CLINICAL TRIAL: NCT00642577
Title: A Randomized, Open Label Study to Compare the Effect of First-line Treatment With Avastin in Combination With Irinotecan + 5-fluorouracil/Folinic Acid, and Irinotecan + 5-fluorouracil/Folinic Acid Alone, on Progression-free Survival in Chinese Patients With Metastatic Colorectal Cancer.
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Chemotherapy in Chinese Patients With Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO20696
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan; Leucovorin; Fluorouracil

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: irinotecan; Drug: leucovorin; Drug: fluorouracil
- 2 (Active Comparator)
  Interventions: Drug: irinotecan; Drug: leucovorin; Drug: fluorouracil

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 5mg/kg iv every 2 weeks
  Arms: 1
Drug: irinotecan — 125mg/m2 iv weekly for 4 weeks of each 6 week cycle
Drug: leucovorin — 20mg/m2 iv weekly for 4 weeks of each 6 week cycle
Drug: fluorouracil — 500mg/m2 iv weekly for 4 weeks of each 6 week cycle

SUMMARY:
This 2 arm study will assess the efficacy and safety of Avastin in combination with irinotecan + 5-fluorouracil/folinic acid, versus irinotecan + fluorouracil/folinic acid alone, as first line treatment in Chinese patients with metastatic colorectal cancer. Patients will be randomized 2:1 to receive 6-weekly cycles of Avastin (5mg/kg iv every 2 weeks) + irinotecan 125mg/m2 iv / leucovorin 20mg/m2 iv / fluorouracil 500mg/m2 iv weekly for 4 weeks, or 6-weekly cycles of irinotecan 125mg/m2 iv / leucovorin 20mg/m2 iv / fluorouracil 500mg/m2 iv weekly for 4 weeks. The anticipated time on study treatment is until disease progression, and the sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* histologically confirmed adenocarcinoma of the colon or rectum, with metastatic disease;
* >=1 measurable lesion;
* ECOG performance status of <=1.

Exclusion Criteria:

* prior systemic therapy for advanced or metastatic disease;
* adjuvant or neo-adjuvant treatment for non-metastatic disease in past 6 months;
* other malignancy within past 5 years, except cured basal cell cancer of skin or cured cancer in situ of cervix;
* clinically significant cardiovascular disease in past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival. | 6 months

SECONDARY OUTCOMES:
Overall response rate, time to response, duration of response, overall survival. | Event driven
AEs, laboratory tests | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- China (9):
  - Beijing
  - Chongqing
  - Guangdong
  - Guangzhou
  - Nanjing
  - Qingdao
  - Shanghai
  - Tianjin
  - Wuhan